CLINICAL TRIAL: NCT00417027
Title: Effect of Manipulation of the Programmed Intermittent Bolus Time Interval and Injection Volume on Total Drug Use for Labor Epidural Analgesia: a Randomized Controlled Trial
Brief Title: Programmed Intermittent Epidural Bolus Time Interval and Injection Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Cynthia Wong, Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524-027
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Results first posted 2011-12-09 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Labor Pain
Keywords: Patient controlled epidural analgesia; Labor analgesia; Epidural analgesia
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2.5 mL bolused every 15 minutes (Active Comparator)
  Interventions: Procedure: Programmed Intermittent Epidural Bolus (PIEB)
- 5ml bolused every 30 minutes (Active Comparator)
  Interventions: Procedure: Programmed Intermittent Epidural Bolus (PIEB)
- 10ml bolused every 60 minutes (Active Comparator)
  Interventions: Procedure: Programmed Intermittent Epidural Bolus (PIEB)

INTERVENTIONS:
Procedure: Programmed Intermittent Epidural Bolus (PIEB) — A commercial pump that can be programmed to administer intermittent boluses and patient controlled boluses does not exist. Two pumps were prepared for each subject with the same epidural solution. One pump was programmed to administer the programmed intermittent epidural bolus(PIEB). The second pump was programmed to administer patient controlled epidural analgesia (PCEA)with a dose of 5 mL delivered with a lockout of every 10 minutes.
  Other Names: Hospira Gemstar infusion pump

SUMMARY:
Studies suggest that administration of maintenance epidural solutions as programmed or automated intermittent boluses, rather than continuous infusions, result in lower bupivacaine consumption, decreased need for manual boluses by the anesthesiologist, and greater patient satisfaction. In this technique, the epidural maintenance dose is administered as a bolus by the infusion pump at regular intervals instead of as a continuous infusion. However, the optimal combination of bolus volume and dosing interval has not been determined. At one end of the spectrum, a small volume and short bolus dose interval will likely behave like a continuous infusion. At the other end of the spectrum, a large volume and long bolus dose interval may lead to an increased incidence of breakthrough pain. The purpose of this randomized, double-blind trial was to determine how manipulation of the programmed intermittent time interval and volume influences total drug use, quality of analgesia, and patient satisfaction during maintenance of labor analgesia. We hypothesized that manipulation of the programmed intermittent bolus time interval and volume during the maintenance of epidural labor analgesia influences total drug use, quality of analgesia and patient satisfaction.

DETAILED DESCRIPTION:
Traditionally, neuraxial labor analgesia was maintained for the duration of labor with manual intermittent bolus injection of anesthetic by the anesthesiologist via an in-dwelling epidural catheter. During the last decade, there has been a transition to maintenance of analgesia with a continuous epidural infusion. Analgesia is maintained with fewer episodes of breakthrough pain and parturient satisfaction is increased. The anesthesiologists' workload is less. More recently, use of patient controlled epidural analgesia (PCEA) has become popular; usually a continuous infusion is supplemented by patient-activated bolus injections.

Studies have compared the intermittent manual epidural bolus technique to continuous infusion, continuous infusion to PCEA without a background infusion, and PCEA with and without a background infusion. Studies vary in the epidural solution local anesthetic mass (volume and concentration), and lock-out intervals. The incidence and intensity of motor blockade is greater with continuous infusion compared to bolus administration of the same concentration/mass local anesthetic per unit time, whether the bolus is administered manually or by PCEA. Consumption of local anesthetic is less with bolus administration (manual or PCEA) compared to continuous infusion. Therefore, lower concentrations of local anesthetic are frequently used for continuous infusions.

Current pump technology supports continuous epidural infusion, PCEA without a background infusion, and PCEA with a background infusion. Current pump technology does not support programmed intermittent bolus administration with or without supplemental PCEA. Further study in this area may motivate pump manufacturers to redesign their pumps to support this type of drug administration.

The purpose of the study is to determine how manipulation of the programmed intermittent time interval and volume influences total drug use, quality of analgesia, and patient satisfaction during maintenance of labor analgesia.

Eligible women were asked to participate shortly after admission to the Labor and Delivery Unit at Prentice Women's Hospital immediately following the routine preanesthetic interview. Informed, written consent was obtained. At the time of request for labor analgesia the cervix was examined and a baseline Visual Analog Scale (VAS) for pain (100 mm unmarked line with the end points labeled "no pain" and "worst pain imaginable") was determined. Labor analgesia was initiated with a routine combined spinal epidural (CSE) technique. The VAS for pain was determined 10 minutes after the intrathecal injection. If the VAS was less than 10 mm, the parturient was randomized (by a computer generated random number table) to one of three programmed intermittent epidural bolus analgesia maintenance techniques: 2.5 mL every 15 minutes, 5 mL every 30 minutes, or 10 mL every 60 minutes. All epidural solutions consisted of bupivacaine 0.0625% with fentanyl 1.95 micrograms/mL. The initial programmed intermittent bolus dose was initiated 30 minutes after the intrathecal injection in all groups.

Programmed intermittent epidural doses were administered via a Hospira Gemstar infusion pump. A commercial pump that can be programmed to administer intermittent boluses and patient controlled boluses does not exist. Thus two pumps were prepared for each subject with the same epidural solution. One pump was programmed to administer the programmed intermittent boluses at a rate of 300 ml/hr at regular intervals. The second pump was programmed to administer the patient's controlled epidural analgesia.

VAS scores for pain were determined every 120 minutes until complete cervical dilation beginning 60 minutes after the intrathecal injection. A modified Bromage score was determined every 120 minutes during the 1st stage of labor (0=no motor paralysis; 1=inability to raise extended leg, but able to move knee and foot; 2=inability to raise extended leg and to move knee, but able to move foot; 3=inability to raise extended leg or to move knee and foot). Sensory threshold to a rigid von Frye filament (pressure applied with the rigid tip until the subject reported feeling pressure at the thoracic dermatome of T12, T10, T7, and T4) was determined bilaterally at initiation of epidural and 3 hours after the intrathecal injection. Epidural infusion was discontinued shortly after delivery. Prior to discharge from the Labor and Delivery Unit the parturient was asked to mark her overall satisfaction with labor analgesia using a 100 mm unmarked line with the left end labeled "not satisfied at all" and the right end labeled "extremely satisfied".

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* nulliparous women
* term gestation (greater than or equal to 37 weeks gestation)
* spontaneous labor or with spontaneous rupture of membranes

Exclusion Criteria:

* Systemic disease (e.g., diabetes mellitus, hypertension, preeclampsia)
* use of chronic analgesic medications
* systemic opioid labor analgesia prior to the initiation of neuraxial labor analgesia
* cervical dilation less than 2cm or greater than 5cm at time of initiation of neuraxial analgesia
* delivery within 90 minutes of intrathecal injection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2006-08; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Wong, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Paech MJ, Pavy TJ, Sims C, Westmore MD, Storey JM, White C. Clinical experience with patient-controlled and staff-administered intermittent bolus epidural analgesia in labour. Anaesth Intensive Care. 1995 Aug;23(4):459-63. doi: 10.1177/0310057X9502300408. PMID 7485937
- [Background] Boutros A, Blary S, Bronchard R, Bonnet F. Comparison of intermittent epidural bolus, continuous epidural infusion and patient controlled-epidural analgesia during labor. Int J Obstet Anesth. 1999 Oct;8(4):236-41. doi: 10.1016/s0959-289x(99)80103-4. PMID 15321117
- [Background] Bogod DG, Rosen M, Rees GA. Extradural infusion of 0.125% bupivacaine at 10 ml h-1 to women during labour. Br J Anaesth. 1987 Mar;59(3):325-30. doi: 10.1093/bja/59.3.325. PMID 3828182
- [Background] Smedstad KG, Morison DH. A comparative study of continuous and intermittent epidural analgesia for labour and delivery. Can J Anaesth. 1988 May;35(3 ( Pt 1)):234-41. doi: 10.1007/BF03010616. PMID 3289768
- [Background] van der Vyver M, Halpern S, Joseph G. Patient-controlled epidural analgesia versus continuous infusion for labour analgesia: a meta-analysis. Br J Anaesth. 2002 Sep;89(3):459-65. doi: 10.1093/bja/aef217. PMID 12402726
- [Background] Paech MJ. Patient-controlled epidural analgesia in labour--is a continuous infusion of benefit? Anaesth Intensive Care. 1992 Feb;20(1):15-20. doi: 10.1177/0310057X9202000103. PMID 1609935
- [Background] Ferrante FM, Rosinia FA, Gordon C, Datta S. The role of continuous background infusions in patient-controlled epidural analgesia for labor and delivery. Anesth Analg. 1994 Jul;79(1):80-4. doi: 10.1213/00000539-199407000-00015. PMID 8010458
- [Background] Boselli E, Debon R, Cimino Y, Rimmele T, Allaouchiche B, Chassard D. Background infusion is not beneficial during labor patient-controlled analgesia with 0.1% ropivacaine plus 0.5 microg/ml sufentanil. Anesthesiology. 2004 Apr;100(4):968-72. doi: 10.1097/00000542-200404000-00030. PMID 15087635
- [Background] Petry J, Vercauteren M, Van Mol I, Van Houwe P, Adriaensen HA. Epidural PCA with bupivacaine 0.125%, sufentanil 0.75 microgram and epinephrine 1/800.000 for labor analgesia: is a background infusion beneficial? Acta Anaesthesiol Belg. 2000;51(3):163-6. PMID 11129615
- [Background] Halonen P, Sarvela J, Saisto T, Soikkeli A, Halmesmaki E, Korttila K. Patient-controlled epidural technique improves analgesia for labor but increases cesarean delivery rate compared with the intermittent bolus technique. Acta Anaesthesiol Scand. 2004 Jul;48(6):732-7. doi: 10.1111/j.0001-5172.2004.00413.x. PMID 15196106
- [Background] Chua SM, Sia AT. Automated intermittent epidural boluses improve analgesia induced by intrathecal fentanyl during labour. Can J Anaesth. 2004 Jun-Jul;51(6):581-5. doi: 10.1007/BF03018402. PMID 15197122
- [Background] Ueda K, Ueda W, Manabe M. A comparative study of sequential epidural bolus technique and continuous epidural infusion. Anesthesiology. 2005 Jul;103(1):126-9. doi: 10.1097/00000542-200507000-00019. PMID 15983464
- [Background] Hogan Q. Distribution of solution in the epidural space: examination by cryomicrotome section. Reg Anesth Pain Med. 2002 Mar-Apr;27(2):150-6. doi: 10.1053/rapm.2002.29748. PMID 11915061
- [Background] Chestnut DH, Owen CL, Bates JN, Ostman LG, Choi WW, Geiger MW. Continuous infusion epidural analgesia during labor: a randomized, double-blind comparison of 0.0625% bupivacaine/0.0002% fentanyl versus 0.125% bupivacaine. Anesthesiology. 1988 May;68(5):754-9. PMID 3285732
- [Background] Li DF, Rees GA, Rosen M. Continuous extradural infusion of 0.0625% or 0.125% bupivacaine for pain relief in primigravid labour. Br J Anaesth. 1985 Mar;57(3):264-70. doi: 10.1093/bja/57.3.264. PMID 3978008
- [Background] Bernard JM, Le Roux D, Vizquel L, Barthe A, Gonnet JM, Aldebert A, Benani RM, Fossat C, Frouin J. Patient-controlled epidural analgesia during labor: the effects of the increase in bolus and lockout interval. Anesth Analg. 2000 Feb;90(2):328-32. doi: 10.1097/00000539-200002000-00017. PMID 10648316
- [Background] Gambling DR, Huber CJ, Berkowitz J, Howell P, Swenerton JE, Ross PL, Crochetiere CT, Pavy TJ. Patient-controlled epidural analgesia in labour: varying bolus dose and lockout interval. Can J Anaesth. 1993 Mar;40(3):211-7. doi: 10.1007/BF03037032. PMID 8467542

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nulliparous women in spontaneous labor were asked to participate shortly after admission to the Labor and Delivery Unit at Prentice Women's Hospital. Immediately following the routine preanesthetic interview, subjects were approached and informed, written consent was obtained.
Groups:
- 2.5 mL Bolused Every 15 Minutes: Laboring women receiving a programmed intermittent epidural bolus of 2.5 ml of bupivacaine 6.25 mg/ml and fentanyl 1.96 mcg/ml every 15 minutes. Patients could request additional 5 ml of the solution via a patient controlled administration every 15 minutes to a maximum of 30ml per hour.
- 5ml Bolused Every 30 Minutes: Laboring women receiving a programmed intermittent epidural bolus of 5 ml of bupivacaine 6.25 mg/ml and fentanyl 1.96 mcg/ml every 30 minutes. Patients could request additional 5 ml of the solution via a patient controlled activation to a maximum of 30 ml per hour.
- 10ml Bolused Every 60 Minutes: Laboring women receiving a programmed intermittent epidural bolus of 10 ml of bupivacaine 6.25 mg/ml and fentanyl 1.96 mcg/ml every 60 minutes. Patients could request additional 5 ml of the solution via a patient controlled activation to a maximum of 30 ml per hour.
Period: Overall Study
Arm/Group | 2.5 mL Bolused Every 15 Minutes | 5ml Bolused Every 30 Minutes | 10ml Bolused Every 60 Minutes
Started | 66 | 65 | 59
Completed | 66 | 60 | 54
Not Completed | 0 | 5 | 5
Not completed — Protocol Violation | 0 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.5 mL Bolused Every 15 Minutes | 5ml Bolused Every 30 Minutes | 10ml Bolused Every 60 Minutes | Total
Number analyzed (Participants) | 66 | 65 | 59 | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 66 | 65 | 59 | 190
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [28 to 33] | 30 [27 to 33] | 31 [28 to 34] | 31 [28 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 65 | 59 | 190
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 66 | 65 | 59 | 190

OUTCOME MEASURES:

1. Primary Outcome: Total Bupivicaine in Milligrams Administered Per Hour of Labor for Analgesia.
Description: Total bupivacaine from epidural solution administered for labor analgesia normalized per hour of labor.
Time Frame: From initiation of labor analgesia until delivery less than 24 hours
Population: per protocal
Measure: Median (Inter-Quartile Range); unit: mg bupivacaine per hour
Arm/Group | 2.5 mL Bolused Every 15 Minutes | 5ml Bolused Every 30 Minutes | 10ml Bolused Every 60 Minutes
Number analyzed (Participants) | 66 | 60 | 54
mg bupivacaine per hour | 11.3 [9.5 to 13.6] | 11.1 [9.2 to 13.3] | 10.3 [8.9 to 11.2]
Statistical Analysis 1: Comparison: 2.5 mL Bolused Every 15 Minutes vs 5ml Bolused Every 30 Minutes; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Bonferroni corrected for 6 comparisons
Statistical Analysis 2: Comparison: 2.5 mL Bolused Every 15 Minutes vs 10ml Bolused Every 60 Minutes; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney) — Bonferroni corrected for 6 comparisons
Statistical Analysis 3: Comparison: 5ml Bolused Every 30 Minutes vs 10ml Bolused Every 60 Minutes; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney) — Bonferroni corrected for 6 comparisons

2. Secondary Outcome: Area Under the Visual Analog Pain Scores (0 to 100mm) Per Hour of Labor Analgesia Curve
Description: The pain burden calculated as the area under the visual analog pain scale (0 to 100 mm) patient self reported assessment of pain. Pain assessment were made at regular intervals during labor and the area under the pain score per time curve was calculated as the pain burden during labor. Greater pain would be indicated by a larger area. Possible range would be 0 for no pain to 100 for severe pain.
Time Frame: Duration of labor analgesia
Population: per protocal
Measure: Median (Inter-Quartile Range); unit: 0 to 100 mm per hour
Arm/Group | 2.5 mL Bolused Every 15 Minutes | 5ml Bolused Every 30 Minutes | 10ml Bolused Every 60 Minutes
Number analyzed (Participants) | 66 | 60 | 54
0 to 100 mm per hour | 15 [6 to 29] | 13 [5 to 26] | 14 [8 to 25]
Statistical Analysis 1: Comparison: 2.5 mL Bolused Every 15 Minutes vs 5ml Bolused Every 30 Minutes vs 10ml Bolused Every 60 Minutes; Test type: Superiority or Other; p = 0.54, Kruskal-Wallis

3. Secondary Outcome: Patient Controlled Bolus Attempts
Description: The number of attempted self administered bolus doses of epidural analgesia solution for control of pain.
Time Frame: Duration of labor analgesia
Population: per protocal
Measure: Mean (Inter-Quartile Range); unit: number of bolus attempts
Arm/Group | 2.5 mL Bolused Every 15 Minutes | 5ml Bolused Every 30 Minutes | 10ml Bolused Every 60 Minutes
Number analyzed (Participants) | 66 | 60 | 54
number of bolus attempts | 10 [3 to 17] | 10 [3 to 17] | 8 [4 to 11]
Statistical Analysis 1: Comparison: 2.5 mL Bolused Every 15 Minutes vs 5ml Bolused Every 30 Minutes vs 10ml Bolused Every 60 Minutes; Test type: Superiority or Other; p = 0.32, Kruskal-Wallis

4. Secondary Outcome: Number of Patient Controlled Bolus Doses of Bupivacaine/Fentanyl Administered
Description: Patient controlled bolus of analgesic solution could be requested by activating a button. Bolus were 5ml of the epidural solution (bupivacaine 6.25mg/ml and fentanyl 1.96mgml). Patient requested administrations were allowed every 10 minutes to a maximum of 30 ml of epidural solution per hour.
Time Frame: Duration of labor analgesia
Population: per protocal
Measure: Mean (Inter-Quartile Range); unit: participants
Arm/Group | 2.5 mL Bolused Every 15 Minutes | 5ml Bolused Every 30 Minutes | 10ml Bolused Every 60 Minutes
Number analyzed (Participants) | 66 | 60 | 54
participants | 7 [3 to 11] | 6 [4 to 10] | 6 [4 to 8]
Statistical Analysis 1: Comparison: 2.5 mL Bolused Every 15 Minutes vs 5ml Bolused Every 30 Minutes vs 10ml Bolused Every 60 Minutes; Test type: Superiority or Other; p = 0.69, Kruskal-Wallis

5. Secondary Outcome: Manual Bolus Doses Administered
Time Frame: Duration of labor analgesia
Measure: Number; unit: participants
Arm/Group | 2.5 mL Bolused Every 15 Minutes | 5ml Bolused Every 30 Minutes | 10ml Bolused Every 60 Minutes
Number analyzed (Participants) | 66 | 60 | 54
participants
  0 doses | 24 | 30 | 27
  1 dose | 23 | 17 | 17
  2 doses | 12 | 11 | 7
  3 doses | 3 | 1 | 1
  4 doses | 4 | 1 | 2
Statistical Analysis 1: Comparison: 2.5 mL Bolused Every 15 Minutes vs 5ml Bolused Every 30 Minutes vs 10ml Bolused Every 60 Minutes; Analysis apply to all rows. Only 1 comparison was made between the groups in distribution of number of bolus doses; Test type: Superiority or Other; p = 0.72, Chi-squared, Corrected — Analysis applies to all rows

6. Secondary Outcome: Highest Thoracic Dermatome Sensory Level to Ice. Higher Levels Are Given by Lower Thoracic Vertebral Number.
Description: Highest level of sensory loss to ice 3 hours after initiation of epidural analgesia. Thoracic dermatomes specify the level at which the nerves exit the spinal column. Higher thoracic spread of analgesia suggests greater dispersion of the epidural solution and may correlate with better analgesia. Higher levels are given by lower thoracic vertebral number. For example dermatome 4 has greater spread than dermatome 5.
Time Frame: 3 hours after initiation of labor analgesia
Measure: Number; unit: participants
Arm/Group | 2.5 mL Bolused Every 15 Minutes | 5ml Bolused Every 30 Minutes | 10ml Bolused Every 60 Minutes
Number analyzed (Participants) | 66 | 60 | 54
participants
  Thoracic dermatome 4 | 6 [7 to 4] | 5 [7 to 5] | 5 [7 to 5]
  Thoracic dermatome 5 | 11 [8 to 6] | 12 [9 to 5] | 9 [9 to 6]
  Thoracic dermatome 6 | 9 | 7 | 8
  Thoracic dermatome 7 | 17 | 14 | 16
  Thoracic dermatome 8 | 10 | 8 | 6
  Thoracic dermatome 9 | 6 | 14 | 10
  Sensory level not tested | 1 | 0 | 0
Statistical Analysis 1: Comparison: 2.5 mL Bolused Every 15 Minutes vs 5ml Bolused Every 30 Minutes vs 10ml Bolused Every 60 Minutes; Test type: Superiority or Other; p = 0.41, Kruskal-Wallis

7. Secondary Outcome: Overall Satisfaction Scores. Higher Scores Represent Greater Satisfaction With Analgesia During Labor and Delivery.
Description: Patient satisfaction with analgesia management during labor and delivery. Scores are 0 to 100 with 0 complete dissatisfaction and 100 complete satisfaction with labor analgesia.
Time Frame: 24 hours following labor analgesia
Population: per protocal
Measure: Median (Inter-Quartile Range); unit: Scores on a scale (0 toi 100)
Arm/Group | 2.5 mL Bolused Every 15 Minutes | 5ml Bolused Every 30 Minutes | 10ml Bolused Every 60 Minutes
Number analyzed (Participants) | 66 | 60 | 54
Scores on a scale (0 toi 100) | 90 [78 to 99] | 94 [80 to 100] | 93 [92 to 98]
Statistical Analysis 1: Comparison: 2.5 mL Bolused Every 15 Minutes vs 5ml Bolused Every 30 Minutes vs 10ml Bolused Every 60 Minutes; Test type: Superiority or Other; p = 0.85, Kruskal-Wallis

ADVERSE EVENTS:
Arm/Group | 2.5 mL Bolused Every 15 Minutes | 5ml Bolused Every 30 Minutes | 10ml Bolused Every 60 Minutes
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/60 | 0/54
Other Adverse Events (participants affected / at risk) | 0/66 | 0/60 | 0/54

LIMITATIONS AND CAVEATS:
No group that received a continuous infusion or PCEA without a background infusion was included. Conclusions are limited to our patient population, drug concentrations, and mode of initiation of labor analgesia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes